CLINICAL TRIAL: NCT02693197
Title: A Phase 1, Two-Part, Open-Label, Parallel-Cohort, Single-Dose Study to Determine the Pharmacokinetics of T-817MA in Adult Subjects With Hepatic Impairment and in Healthy Adult Subjects
Brief Title: PK Study of T-817 in Subjects With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FUJIFILM Toyama Chemical Co., Ltd. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: T817MAUS113
Record Dates: First submitted 2016-01-26; First posted 2016-02-26 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-05

CONDITIONS: Healthy; Hepatic Impairment
Keywords: Hepatic Impairment
MeSH Terms: interventions — 1-(3-(2-(1-benzothiophen-5-yl) ethoxy) propyl)-3-azetidinol maleate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1:T-817MA (Experimental): Mild hepatic impairment subjects
  Interventions: Drug: T-817MA
- Cohort 2:T-817MA (Experimental): Healthy subjects matched to subjects in Cohort 1
  Interventions: Drug: T-817MA
- Cohort 3:T-817MA (Experimental): Moderate hepatic impairment subjects
  Interventions: Drug: T-817MA
- Cohort 4:T-817MA (Experimental): Healthy subjects matched to subjects in Cohort 3
  Interventions: Drug: T-817MA
- Cohort 5 :T-817MA (Experimental): Severe hepatic impairment subjects
  Interventions: Drug: T-817MA
- Cohort 6:T-817MA (Experimental): Healthy subjects matched to subjects in Cohort 5
  Interventions: Drug: T-817MA

INTERVENTIONS:
Drug: T-817MA — A single oral dose of 448 mg

SUMMARY:
The primary objective is to determine the single-dose pharmacokinetics (PK) of T-817 and T-817M5 (metabolite of T-817) in subjects with mild, moderate or severe hepatic impairment compared to matched healthy control subjects.

The secondary objective is to determine the safety and tolerability of single-dose T -817MA (Maleate salt of T-817) in subjects with mild, moderate or severe hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

For subjects with mild, moderate or severe hepatic impairment

1. Adult male or female, 18 - 75 years of age
2. Must weigh at least 50 kg and have a body mass index (BMI) ≥ 18.5 and ≤ 40.0 kg/m2
3. Have mild, moderate or severe defined by Child-Pugh classification hepatic impairment

For Matched Healthy Control Subjects Healthy adult male or female subjects will be matched 1:1 to a specific subject in the mild, moderate, or severe hepatic impairment cohort based upon age, weight, gender, and smoking status

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI.
3. History or presence of hypersensitivity or idiosyncratic reaction to the study drug, related compounds, or inactive ingredients.
4. Female subjects who are pregnant or lactating.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations | 8 days
Area under the plasma concentration time curve (AUC) | 8 days
Maximum observed plasma concentration (Cmax) | 8 days
Time to reach the maximum observed plasma concentration (tmax) | 8 days
Apparent terminal elimination rate constant | 8 days
Apparent terminal elimination half-life (t½) | 8 days
Apparent total plasma clearance of unbound drug after oral (extravascular) administration (CL/F) | 8 days
Apparent volume of distribution during the terminal elimination phase after oral (extravascular) administration (Vd/F) | 8 days
Metabolite to parent ratio (MPR) | 8 days

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 8days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Preston, M.D., Principal Investigator — University of Miami; Thomas Marbury, M.D., Principal Investigator — Orlando Clinical Research Center
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida